CLINICAL TRIAL: NCT05706012
Title: Long-term Antithrombotic Management of Acute Mesenteric Ischaemia: Case-based Survey
Brief Title: Antithrombotic Management of Acute Mesenteric Ischaemia
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s67503
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-11

CONDITIONS: Acute Mesenteric Ischemia; Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastro-enterologists and anticoagulation specialists: An online survey will be sent to question current clinical practice in long-term antithrombotic management of AMI in SBS patients.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Online survey questioning the current clinical practice on long-term antithrombotic management of AMI in SBS patients

SUMMARY:
Guidelines on the acute and long-term pharmacological treatment of acute mesenteric ischaemia (AMI) recommend the use of thrombolytic, antiplatelet or anticoagulant therapy depending on the aetiology of AMI and the use of stenting but only few details are given on the choice of the drug, dose and duration of treatment. Besides, recommendations are mainly based on data on coronary, cerebral and other peripheral artery diseases and do also not take into account the altered drug absorption in patients with short bowel syndrome, in which AMI can result.This case-based survey will inform us on the current international clinical practice of long-term antithrombotic management of AMI.

ELIGIBILITY:
Inclusion Criteria:

* gastro-enterologist or cardiologist with expertise in treating SBS patients resulting from AMI

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: international gastro-enterologists an cardiologists
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Type of antithrombotic therapy | April 2023
  Overview of the type of long-term antithrombotic therapy that is prescribed in SBS patients with AMI, depending on the anatomy of the gastrointestinal tract, the aetiology of AMI and whether or not revascularisation of the occluding blood vessel has been performed

SECONDARY OUTCOMES:
Duration of antithrombotic therapy | April 2023
  Overview of the duration of long-term antithrombotic therapy in SBS patients with AMI depending on the anatomy of the gastrointestinal tract, the aetiology of AMI and whether or not revascularisation of the occluding blood vessel has been performed.
Initial dose of antithrombotic therapy | April 2023
  Overview of the initial dose of long-term antithrombotic therapy in SBS patients with AMI depending on the anatomy of the gastrointestinal tract, the aetiology of AMI and whether or not revascularisation of the occluding blood vessel has been performed.
Dose adjustments of antithrombotic therapy | April 2023
  Overview of any dose adjustments of long-term antithrombotic therapy in SBS patients with AMI depending on the anatomy of the gastrointestinal tract, the aetiology of AMI and whether or not revascularisation of the occluding blood vessel has been performed.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
no IPD will be shared with other researchers